CLINICAL TRIAL: NCT01003951
Title: Acupuncture for the Treatment of Chronic Lymphedema: A Feasibility Study
Brief Title: Acupuncture for the Treatment of Chronic Lymphedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-136
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer; Lymphedema
Keywords: Lymphedema; Acupuncture; 09-136
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Acupuncture Therapy

ARMS (1):
- Acupuncture (Experimental): Each patient will receive two acupuncture treatments each week for four consecutive weeks. At the end of four weeks, the intervention will be complete.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture treatments will be given at the Integrative Medicine Outpatient Center, if needed in particular cases, at the MSKCC Breast Center. Each treatment is 30-40 minutes in duration. Each patient will receive two acupuncture treatments each week for four consecutive weeks.
  Before and after each treatment, the circumference of the patient's upper arm, and forearm will be measured in both the affected and unaffected arms. The greater difference between affected and unaffected arms (either the forearm or the upper arm) for each patient will be used for outcome assessment. Photographs of the patient's affected and unaffected arms before and after each treatment will be taken to provide visual documentation of status. The patient's face will not appear in the photographs. Blood draws will be performed from the unaffected arm in serum collection tubes and will be performed within 1 week of starting acupuncture and within 1 week of completion of the 4 week protocol.

SUMMARY:
Lymphedema is an accumulation of lymphatic fluid in the tissues that causes swelling, most often in the arms and/or legs, and occasionally in other parts of the body. Lymphedema can occur when lymph vessels are damaged or lymph nodes are removed. Lymphedema can develop right after breast cancer treatment or weeks, months, or even years later. For many people, available treatments for lymphedema are not effective. Recent evidence suggests that acupuncture may help reduce the symptoms of lymphedema. The purpose of this study is to determine the effects of acupuncture on chronic lymphedema. This study will look further at whether acupuncture can reduce lymphedema and help us to understand immune changes that may be associated with improvements in lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 or older willing to sign consent.
* Lymphedema in an arm as a result of surgery, chemotherapy, and/or radiation therapy for breast cancer per Breast surgeon or medical oncologist.
* Patients must have received a clinical diagnosis of lymphedema for at least 6 months and no more than 5 years after diagnosis of chronic lymphedema.
* The affected arm must be >2cm larger than the unaffected arm; this is the standard diagnosis and the one used in the MSKCC studies cited above. The standard measurement techniques will be applied 20.

Exclusion Criteria:

* Previous acupuncture treatment for lymphedema
* Diuretic use
* History of primary (congenital) lymphedema
* Metastatic cancer
* History of autoimmune disorder (including lupus, rheumatoid arthritis, systemic sclerosis)
* History of other fibroproliferative disorder including cirrhosis, pulmonary fibrosis, kidney fibrosis, systemic sclerosis/scleroderma
* Current treatment with corticosteroids
* Treatment with myelosuppressive or stimulatory drugs within 6 months of enrollment
* History of bone marrow transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To obtain preliminary evidence of the effects of acupuncture on chronic lymphedema due to breast cancer treatment. | twice weekly for four consecutive weeks and will be followed for an additional 6 months

SECONDARY OUTCOMES:
To further evaluate the safety of acupuncture in this setting. | 6 months to record any side effects that may occur post-treatment
To obtain preliminary evidence of systemic immune changes that occur after acupuncture treatment of lymphedema. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Barrie Cassileth, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Cassileth BR, Van Zee KJ, Yeung KS, Coleton MI, Cohen S, Chan YH, Vickers AJ, Sjoberg DD, Hudis CA. Acupuncture in the treatment of upper-limb lymphedema: results of a pilot study. Cancer. 2013 Jul 1;119(13):2455-61. doi: 10.1002/cncr.28093. Epub 2013 Apr 10. PMID 23576267
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm